CLINICAL TRIAL: NCT01949441
Title: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled Parallel-Group Study to Assess the Tolerability of ToleroMune House Dust Mite in Subjects With Controlled Asthma and House Dust Mite-Induced Rhinoconjunctivitis
Brief Title: ToleroMune House Dust Mite (HDM) Tolerability Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH004
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Rhinoconjunctivitis
Keywords: HDM Allergy; Rhinoconjunctivitis; Immunotherapy; ToleroMune HDM

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ToleroMune HDM (Experimental)
  Interventions: Biological: ToleroMune HDM
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ToleroMune HDM — Intradermal injection 1 x 4 administrations 4 weeks apart
  Arms: ToleroMune HDM
Biological: Placebo — Intradermal injection 1 x 4 administrations 4 weeks apart
  Arms: Placebo

SUMMARY:
House Dust Mites (HDMs) are arachnids that infest bedding, carpet, upholstered furniture and fabric. Like many other allergens, exposure to HDMA in sensitised patients is associated with poorer lung function, greater medication requirements and more asthma symptoms as well as chronic rhinosinusitis symptoms. In contrast to other allergens, there is evidence that HDMA leads to the development of asthma, in addition to exacerbating pre-existing asthma in HDM-sensitised patients.

ToleroMune House Dust Mite (TM-HDM), a combination of seven Synthetic Peptide Immuno-Regulatory Epitopes, is being developed for the treatment of HDM allergy.

This study to assess the tolerability of ToleroMune House Dust Mite in subjects with controlled asthma and house dust mite-induced rhinoconjunctivitis.

DETAILED DESCRIPTION:
A multi-centre, randomised, double-blind, placebo-controlled, parallel-group, multiple dose study to evaluate the tolerability of four intradermal doses of TM-HDM in subjects with controlled asthma and HDM-induced rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years.
* Asthma controlled by Step 1 or Step 2 treatment as defined by GINA in the four weeks prior to randomisation.
* Asthma controlled by Step 1 or Step 2 treatment as defined by GINA in the four weeks prior to randomisation.
* No change in asthma controller treatment (dose, frequency) in the four weeks prior to randomisation.
* A reliable history consistent with rhinoconjunctivitis on exposure to HDM for at least 1 year that has required symptomatic treatment on at least one occasion during the year prior to randomisation
* Positive skin prick test to Dermatophagoides pteronyssinus with an average wheal diameter at least 5 mm larger than that produced by the negative control.
* ImmunoCAP® Dermatophagoides pteronyssinus-specific Immunoglobulin E ≥ 0.35 kU/L.

Exclusion Criteria:

* History of life-threatening asthma
* Asthma exacerbation in the 12 weeks prior to randomisation
* Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) < 80 % of predicted, regardless of the cause.
* Post-bronchodilator FEV1/Forced Vital Capacity ratio of < 0.7.
* Concurrent respiratory disease that would confound study participation or affect subject safety.
* Non-HDM allergy that may significantly interfere with the results of this study.

  7. Previous immunotherapy treatment with any HDM allergen for more than 1 month within 5 years prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 19 Weeks

SECONDARY OUTCOMES:
FEV1 and FVC | Up to 19 Weeks
Peak Expiratory Flow Rate | Up to 19 Weeks
VAS Breathlessness | Up to 19 weeks
Asthma Exacerbations | Up to 19 weeks
Systemic Allergic Reactions | Up to 19 Weeks
Injection Site Examinations | Up to 19 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Topstone Research, Toronto, Ontario, Canada